CLINICAL TRIAL: NCT07094295
Title: Association of Perioperative Blood Transfusion With Increased One-year Mortality After Surgery: a Retrospective Propensity Score-Matched Cohort Study
Brief Title: Perioperative Blood Transfusion and Increased One-year Mortality
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Wen-bin Lu, MD, Principal Investigator, Changhai Hospital
Other Study IDs: PBTOM
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mortality, Perioperative Blood Transfusion, Propensity Score, Retrospective Study, Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PBT group: Patients in PBT group received red blood cell concentrate units during surgery and up to one month postoperatively.
  Interventions: Other: perioperative blood transfusion
- No-PBT group: Patients in No-PBT group did not receive red blood cell concentrate units during surgery and up to one month postoperatively.

INTERVENTIONS:
Other: perioperative blood transfusion — The PBT group received the red blood cell concentrate units during surgery and up to one month postoperatively.
  Groups: PBT group

SUMMARY:
The goal of this retrospective observational study is to explore the association of perioperative blood transfusion with increased one-year mortality in patients undergoing surgeries. The main question it aims to answer perioperative blood transfusion is associated with increased one-year mortality across various surgical settings. We will retrospectively collect the clinical data (including one-year mortality) in patients with perioperative blood transfusion or not and analysis the association between perioperative blood transfusion and one-year mortality after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Patients undergoing first-time cardiothoracic surgery, orthopedics, obstetrics and gynecology, general surgery, otolaryngology, hand surgery, neurosurgery, colorectal surgery, urology, plastic surgery, and oral and maxillofacial surgery were included.

Exclusion Criteria:

* Patients with missing values for the American Society of Anesthesiologists (ASA) physical status, revised cardiac risk index (RCRI), degree of preoperative anemia, kidney disease, or race were excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent surgery at Singapore General Hospital between 1 January 2012 and 31 October 2016
Sampling Method: Non-Probability Sample
Enrollment: 97443 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
one-year mortality after surgery | one year after surgery